CLINICAL TRIAL: NCT03770325
Title: Effect of Berberine on Cardiovascular Disease Risk Factors: a Mechanistic Randomized Controlled Trial
Brief Title: A Mechanistic Randomized Controlled Trial on the Cardiovascular Effect of Berberine
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Food and Health Bureau, Hong Kong (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 15162621
Record Dates: First submitted 2018-12-03; First posted 2018-12-10 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Cardiovascular Risk Factor
MeSH Terms: interventions — Berberine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Berberine (Experimental): berberine (500 mg orally twice a day)
  Interventions: Drug: Berberine
- Placebo (Placebo Comparator): placebo (500 mg orally twice a day)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Berberine — Purified berberine (500 mg orally twice a day) in tablets for 12 weeks
  Arms: Berberine
Drug: Placebo — Placebo tablets, prepared with the same appearance, for 12 weeks
  Arms: Placebo

SUMMARY:
Berberine is extracted from Coptis (Huanglian) and Phellodendron Chinese (Huangbai), to make into berberine tablets.1 Recent studies have shown that berberine has beneficial effects on cardiovascular disease (CVD) risk factors,1,2 such as lowering the risk of hyperlipidemia, diabetes, and hypertension.1 In a comprehensive systematic review and meta-analysis of 27 randomized controlled trials (RCTs), berberine effectively reduced low density lipoprotein cholesterol (LDL-c) (-0.65 mmol/L, 95% confidence interval (CI) -0.75 to -0.56), triglycerides (TG) (-0.39 mmol/L, 95% CI -0.59 to -0.19), total cholesterol (TC) (-0.66 mmol/L, 95% CI -1.02 to -0.31) and increased high density lipoprotein cholesterol (HDL-c) (0.07mmol/L, 95% CI 0.04 to 0.1).1 Notably, no serious adverse event has been reported in these trials,1 suggesting a good tolerability of berberine. The mechanism by which berberine exerts a protective role in atherosclerosis is unclear. Protoberberines have been identified as a new inhibitor of AKR1C3, an enzyme responsible for the regulation of steroid hormone action.3 The investigators propose to examine the effects of berberine on a set of well-established CVD risk factors including lipids, systolic and diastolic blood pressure, coagulation factors, adiposity, fasting glucose, insulin, and liver function, as well as to examine potential mediation via testosterone and/or sex hormone binding globulin using a mechanistic, randomized, double-blind, placebo-controlled trial in Chinese men with hyperlipidemia.

DETAILED DESCRIPTION:
Objectives: to assess the effect of berberine on a set of well-established CVD risk factors, including lipids, systolic and diastolic blood pressure, coagulation factors, fasting glucose, insulin, adiposity (body mass index (BMI) and waist-hip ratio (WHR)) and the mediation via testosterone and/or sex hormone binding globulin using a mechanistic, parallel RCT.

Study design: a mechanistic, randomized, double-blind, placebo-controlled, parallel trial in 84 Chinese men in Hong Kong.

Interventions: the eligible participants will be randomized to take berberine (500 mg orally twice a day) or placebo for 12 weeks. Blood samples will be taken at baseline, 8-week and 12-week intervention.

Data analysis and expected results: the investigators will use an intention to treat analysis, with multiple imputation for missing data. The investigators will compare the baseline characteristics of participants in the two arms using analysis of variance. The investigators will assess the effects of berberine on changes in CVD risk factors using analysis of variance, and the mediation using causal mediation analysis. Compared to the placebo group, the participants receiving berberine are expected to have lower burden of cardiovascular disease risk factors at the end of the intervention. These effects may be mediated or partly mediated by lowering testosterone.

ELIGIBILITY:
Inclusion Criteria:

* Men, who are

  1. aged 20 to 65 years
  2. of Chinese ethnicity
  3. with hyperlipidemia, defined as TG greater than 150 mg/dl (1.70 mmol/L), TC greater than 200 mg/dl (5.16 mmol/L), and/or LDL-c greater than 100 mg/dl (2.58 mmol/L)
  4. willing to make return visits
  5. not currently receiving hormone replacement therapy, such as testosterone replacement therapy, in the past 12 months
  6. not currently taking berberine or traditional Chinese medicine that contains berberine, in the past 1 month
  7. free of any congenital diseases, including familial hypercholesterolemia
  8. free of any infectious diseases, e.g. seasonal influenza
  9. free of anemia and glucose-6-phosphate dehydrogenase deficiency
  10. with no history of any chronic diseases including ischemic heart disease, myocardial infarction (heart attack), stroke, diabetes, cancer, liver/renal dysfunction, and gastrointestinal disorders.

Exclusion Criteria:

* All women, and men, who did not meet the aforementioned inclusion criteria, and/or unable or unwilling to provide consent

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
lipid profile | change from baseline lipid profile at 8 weeks
  LDL-cholesterol, HDL-cholesterol, triglycerides and total cholesterol in mmol/L
lipid profile | change from baseline lipid profile at 12 weeks
  LDL-cholesterol, HDL-cholesterol, triglycerides and total cholesterol in mmol/L
blood pressure | change from baseline blood pressure at 8 weeks
  systolic blood pressure and diastolic blood pressure in mmHg
blood pressure | change from baseline blood pressure at 12 weeks
  systolic blood pressure and diastolic blood pressure in mmHg
thromboxane A2 | change from baseline thromboxane A2 at 8 weeks
  thromboxane A2 in mmol/L
thromboxane A2 | change from baseline thromboxane A2 at 12 weeks
  thromboxane A2 in mmol/L
testosterone | change from baseline testosterone at 8 weeks
  testosterone in mmol/L
testosterone | change from baseline testosterone at 12 weeks
  testosterone in mmol/L
body mass index (BMI) | change from baseline body mass index at 8 weeks
  weight and height will be combined to report BMI in kg/m^2
body mass index (BMI) | change from baseline body mass index at 12 weeks
  weight and height will be combined to report BMI in kg/m^2
waist hip ratio | change from baseline waist hip ratio at 8 weeks
  waist circumstance and hip circumstance will be combined to report waist hip ratio
waist hip ratio | change from baseline waist hip ratio at 12 weeks
  waist circumstance and hip circumstance will be combined to report waist hip ratio
fasting glucose | change from baseline fasting glucose at 8 weeks
  fasting glucose in mmol/L
fasting glucose | change from baseline fasting glucose at 12 weeks
  fasting glucose in mmol/L
fasting insulin | change from baseline fasting insulin at 8 weeks
  fasting insulin in mmol/L
fasting insulin | change from baseline fasting insulin at 12 weeks
  fasting insulin in mmol/L
liver function | change from baseline fasting insulin at 8 weeks
  Alanine transaminase (ALT), Aspartate aminotransferase (AST), Alkaline phosphatase (ALP), total bilirubin, Gamma-glutamyltransferase, total protein and albumin in mmol/L
liver function | change from baseline fasting insulin at 12 weeks
  Alanine transaminase (ALT), Aspartate aminotransferase (AST), Alkaline phosphatase (ALP), total bilirubin, Gamma-glutamyltransferase, total protein and albumin in mmol/L
sex hormone binding globulin (SHBG) | change from baseline SHBG at 8 weeks
  SHBG in nmol/L
sex hormone binding globulin (SHBG) | change from baseline SHBG at 12 weeks
  SHBG in nmol/L
thrombin time | change from baseline thrombin time at 8 weeks
  thrombin time in sec
thrombin time | change from baseline thrombin time at 12 weeks
  thrombin time in sec

CONTACTS AND LOCATIONS:
Overall Officials: Jie Zhao, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Li Ka Shing Faculty of Medicine, Hong Kong, Hong Kong

REFERENCES:
- [Background] Lan J, Zhao Y, Dong F, Yan Z, Zheng W, Fan J, Sun G. Meta-analysis of the effect and safety of berberine in the treatment of type 2 diabetes mellitus, hyperlipemia and hypertension. J Ethnopharmacol. 2015 Feb 23;161:69-81. doi: 10.1016/j.jep.2014.09.049. Epub 2014 Dec 10. PMID 25498346
- [Background] Imanshahidi M, Hosseinzadeh H. Pharmacological and therapeutic effects of Berberis vulgaris and its active constituent, berberine. Phytother Res. 2008 Aug;22(8):999-1012. doi: 10.1002/ptr.2399. PMID 18618524
- [Background] Skarydova L, Hofman J, Chlebek J, Havrankova J, Kosanova K, Skarka A, Hostalkova A, Plucha T, Cahlikova L, Wsol V. Isoquinoline alkaloids as a novel type of AKR1C3 inhibitors. J Steroid Biochem Mol Biol. 2014 Sep;143:250-8. doi: 10.1016/j.jsbmb.2014.04.005. Epub 2014 Apr 24. PMID 24769118